CLINICAL TRIAL: NCT06235710
Title: Prevalence of Musculoskeletal Complaints in Nursing Home Residents
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL84320.068.23
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-05

CONDITIONS: Rheumatoid Arthritis; Rheumatic Diseases; Musculoskeletal Diseases; Musculoskeletal Diseases or Conditions; Gout; Degenerative Joint Disease; Orthopedic Disorder; Arthritis; Polyarthritis; Musculoskeletal Pain; Arthrosis
Keywords: Rheumatic and musculoskeletal diseases; Prevalence; Nursing home residents
MeSH Terms: conditions — Arthritis, Rheumatoid; Rheumatic Diseases; Musculoskeletal Diseases; Gout; Joint Diseases; Arthritis; Musculoskeletal Pain; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Nursing home residents without dementia: * Mentally competent nursing home resident ≥ 65 years;
  * No diagnosis of dementia (major neurocognitive disorder according to DSM-5 criteria);
  * The nursing home resident provides informed consent to participate in the study.
  In this study, nursing home residents all undergo a physical examination of the musculoskeletal system.
  In addition:
  - In group 1: nursing home residents provide an answer on 3 non-incriminating questions (assessment general health, severity of joint complaints and pain in general).
- Group 2: Nursing home residents with dementia: * Nursing home resident with dementia (major neurocognitive disorder according to DSM-5 criteria) ≥ 65 years;
  * The legal representative of the nursing home resident provides informed consent to participate in the study.
  In this study, nursing home residents all undergo a physical examination of the musculoskeletal system.
  In addition:
  In group 2: if possible, provide an answer on 1 non-incriminating question (severity of joint complaints). If the nursing home resident cannot answer this question (reliably), we use the Pain Assessment Checklist for Seniors with Severe Dementia (PACSLAC-D).

SUMMARY:
The goal of this observational study is to investigate the prevalence of joint complaints in nursing home residents with and without dementia.

Primary objective: Number of tender or swollen joints.

Secondary objectives:

1. Only when it is possible for the nursing home resident to provide us this information: how nursing home residents themselves assess the severity of their joint complaints that day (at that time). If the nursing home resident cannot answer this question (reliably), the investigators use the Pain Assessment Checklist for Seniors with Severe Dementia (PACSLAC-D).
2. Investigate mobility limitations among nursing home residents.
3. To understand whether an accurate (differential) diagnosis for the joint complaints is reported in the electronic files.

During the study, a standard physical examination of the musculoskeletal system will performed. Nursing home residents allocated in group 1 (no dementia) also provide an answer on 3 non-incriminating questions (severity of joint complaints, pain in general and general health).

Nursing home residents allocated in group 2 (dementia) answer, if possible, 1 non-incriminating question (pain in joints at that moment). These question(s) and the physical examination are also widely used in daily clinical practice. No further incriminating questions or questionnaires will be administered. If the nursing home resident cannot answer this question (reliably), the investigators use the PACSLAC-D.

DETAILED DESCRIPTION:
Rationale: In older people, alterations in symptom presentation of Rheumatic and Musculoskeletal Diseases (RMDs), objective signs of disease and presence of co-morbidities can pose diagnostic problems and contribute to both over- and undertreatment of RMDs. This is especially the case in nursing home residents. Insight into the prevalence of RMDs and RMD related pain in nursing home residents is currently low. Early recognition and tailored treatment of RMDs may however prevent further loss of mobility, improve quality of life and the quality of medical care of nursing homes residents.

Objectives:

Primary objective: to investigate the prevalence of joint complaints in nursing home residents with and without dementia (major neurocognitive disorder according to DSM-5 criteria). Our definition of joint complaints is: number of tender and / or swollen joints.

Secondary objectives:

1. Only when it is possible for the nursing home resident to provide us this information: how nursing home residents themselves assess the severity of their joint complaints that day (at that time). If the nursing home resident cannot answer this question (reliably), the investigators use the Pain Assessment Checklist for Seniors with Severe Dementia (PACSLAC-D).
2. Investigate mobility limitations among nursing home residents.
3. To understand whether an accurate (differential) diagnosis for the joint complaints is reported in the electronic files.

Study design: observational study, data collection in nursing home residents. Study population: In total, 50 nursing home residents without dementia (group 1) and 50 nursing home residents with dementia (group 2), ≥ 65 years of age, will be included.

Main study parameters/endpoints: During the study, a standard physical examination of the musculoskeletal system will performed. Nursing home residents allocated in group 1 also provide an answer on 3 non-incriminating questions (severity of joint complaints, pain in general and general health).

Nursing home residents allocated in group 2 answer, if possible, 1 non-incriminating question (pain in joints at that moment). These question(s) and the physical examination are also widely used in daily clinical practice. No further incriminating questions or questionnaires will be administered. If the nursing home resident cannot answer this question (reliably), the investigators use the PACSLAC-D.

Expected outcomes and endpoints:

Primary outcome: number of nursing home residents, with and without dementia, with joint complaints; average number of painful and number of swollen joints.

Secondary outcomes:

1. The average level of joint pain on that day, determined by a VAS scale (0-10, 0 no joint pain; 10 a lot of joint pain). If the nursing home resident cannot answer this question (reliably), result of the PACSLAC-D.
2. Amount and severity of mobility limitations among nursing home residents (% independent / % cane or walker / % wheelchair / % bedridden / % combination).
3. More information on how accurately RMDs are reported in the electronic patient files of the nursing home resident. Discrepancy percentage between findings musculoskeletal physical examination versus previously recorded findings in the electronic patient files.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All measurements are performed by trained clinician-researchers using standardized protocols. All participants need to undergo a physical examination of the musculoskeletal system and answer 1-3 questions. No study-specific blood samples are collected during this study. However, in nursing home residents who are under the care of the Cicero care group, a standard blood sample is taken once to twice a year. The laboratory result of the blood sample (C-reactive protein) within a maximum of 3 months before or after the physical examination is also included in this study.

With regard to participation risks and benefits:

Nursing home residents with and without dementia differ significantly from community-dwelling older adults. Multimorbidity, geriatric syndromes and continuous need for complex care are far more common in nursing home residents. Therefore, recommendations on the diagnosis and management of RMDs and musculoskeletal pain in community-dwelling older adults cannot simply be adopted. Nursing home residents with dementia also clearly differ from residents without dementia. As an example: musculoskeletal symptoms such as rigidity, balance problems or a shuffling gait due to unrelieved pain because of arthritis, might be more common in nursing home residents with dementia. For this reason, it is important that nursing home residents with dementia are also included in our study.

Abnormalities during physical examination of potential clinical importance will always be discussed with the nursing home resident / legal representative and their elderly care physician. Awareness of normally unknown pathology may affect a person's perception of his/her own health condition negatively. On the other hand, detection of for instance arthritis has potentially favourable effects on disease progression and may enable early intervention.

Part of the study participants, i.e. those with dementia in group 2, are mentally incompetent / incapacitated. In the event of clear protest / resistance from a nursing home resident, the physical examination will be discontinued. To determine whether there is any protest / resistance, a person who knows the nursing home resident well is always present during the physical examination. This can be the elderly care physician or a nurse. This person has a good understanding of the pattern of habits and behaviours appropriate to that person.

ELIGIBILITY:
Inclusion criteria, group 1:

* Mentally competent nursing home resident ≥ 65 years;
* No diagnosis of dementia (major neurocognitive disorder according to DSM-5 criteria);
* The nursing home resident provides informed consent to participate in the study.

Inclusion criteria, group 2:

* Nursing home resident with dementia (major neurocognitive disorder according to DSM-5 criteria) ≥ 65 years;
* The legal representative of the nursing home resident provides informed consent to participate in the study.

Exclusion criteria, group 1:

* Diagnosis dementia;
* Life expectancy < 2 weeks (definition terminal nursing home resident). Exclusion criteria, group 2
* Life expectancy < 2 weeks (definition terminal nursing home resident).
* If, on the basis of an already known pattern of behaviour, it is expected that the potential participant will resist the proposed research (anticipated behaviour).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: In total, 50 nursing home residents without dementia (group 1) and 50 nursing home residents with dementia (group 2), ≥ 65 years of age, will be included.
  In the Cicero Zorggroep nursing homes, residents are comparable to those living in other nursing homes in the Netherlands. They undergo the same assessment and screening (in the case of psychogeriatric care: mainly ZZP 5, and in somatic care mainly ZZP 6). Within Cicero, there are no specialized departments (e.g., for Parkinson's disease or young dementia patients), so each department consists of a representative cross-section of nursing home residents. In our study, we do not differentiate between subgroups, except for gender and the presence of dementia.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of joint complaints in nursing home residents with and without dementia. | Day 1
  Our definition of joint complaints is: number of tender and / or swollen joints.

SECONDARY OUTCOMES:
The severity of their joint complaints that day. | Day 1
  the average level of joint pain on that day, determined by a VAS scale (0-10, 0 no joint pain; 10 a lot of joint pain). If the nursing home resident cannot answer this question (reliably), we use the Pain Assessment Checklist for Seniors with Severe Dementia (PACSLAC-D).
Amount and severity of mobility limitations among nursing home residents. | Day 1
  % independent / % cane or walker / % wheelchair / % bedridden / % combination
Information on whether an accurate (differential) diagnosis for the joint complaints is reported in the electronic files. | Day 1
  Discrepancy percentage between findings of the musculoskeletal physical examination versus previously recorded findings in the electronic files of the nursing home resident.

OTHER OUTCOMES:
Additional information collected from the electronic patient files. | Day 1
  * General information: age (years), gender, smoking and alcohol consumption.
  * History, co-morbidity and previous operations. Special attention to RMDs, including fractures.
  * Charlson comorbidity index.
  * Only for group 2: type of dementia.
  * Current medication use.
  * Weight (kg), height (cm), blood pressure (mmHg) and heart rate.
  * Fall frequency (falls/year)
  * Information on activities of Daily Living (ADL) extracted from the care plan, with information about getting in and out of bed, dressing and undressing, eating and drinking.

CONTACTS AND LOCATIONS:
Overall Officials: Marloes van Onna, MD; PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Cicero Zorggroep, Brunssum, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
I have not yet chosen a metadata scheme. I will make the following endproducts avaiable for further research and verification: raw data, data documentation, documentation of the research process, including documentation of all participants and syntaxes.

REFERENCES:
- [Background] Abell JE, Hootman JM, Helmick CG. Prevalence and impact of arthritis among nursing home residents. Ann Rheum Dis. 2004 May;63(5):591-4. doi: 10.1136/ard.2003.015479. PMID 15082494
- [Background] Achterberg WP, Pot AM, Scherder EJ, Ribbe MW. Pain in the nursing home: assessment and treatment on different types of care wards. J Pain Symptom Manage. 2007 Nov;34(5):480-7. doi: 10.1016/j.jpainsymman.2006.12.017. Epub 2007 Jul 5. PMID 17616332
- [Background] J. Alaba, E. Arriola, Pain prevalence among the elderly in care homes. Spanish, Revista de la Sociedad Espanola del Dolor 16(6) (2009) 344-351.
- [Background] Al-Momani M, Al-Momani F, Alghadir AH, Alharethy S, Gabr SA. Factors related to gait and balance deficits in older adults. Clin Interv Aging. 2016 Aug 9;11:1043-9. doi: 10.2147/CIA.S112282. eCollection 2016. PMID 27570449
- [Background] Albertsen N, Olsen TM, Sommer TG, Prischl A, Kallerup H, Andersen S. Who lives in care homes in Greenland? A nationwide survey of demographics, functional level, medication use and comorbidities. BMC Geriatr. 2021 Sep 18;21(1):500. doi: 10.1186/s12877-021-02442-0. PMID 34536989
- [Background] Algameel M. Patterns of medication use and adherence to medications among residents in the elderly homes. Pak J Med Sci. 2020 May-Jun;36(4):729-734. doi: 10.12669/pjms.36.4.1923. PMID 32494264
- [Background] Altiparmak S, Altiparmak O. Drug-using behaviors of the elderly living in nursing homes and community-dwellings in Manisa, Turkey. Arch Gerontol Geriatr. 2012 Mar-Apr;54(2):e242-8. doi: 10.1016/j.archger.2011.09.014. Epub 2011 Oct 29. PMID 22037245
- [Background] Bekhet AK, Zauszniewski JA. Chronic conditions in elders in assisted living facilities: associations with daily functioning, self-assessed health, and depressive symptoms. Arch Psychiatr Nurs. 2014 Dec;28(6):399-404. doi: 10.1016/j.apnu.2014.08.013. Epub 2014 Sep 3. PMID 25457691
- [Background] Black BS, Finucane T, Baker A, Loreck D, Blass D, Fogarty L, Phillips H, Hovanec L, Steele C, Rabins PV. Health problems and correlates of pain in nursing home residents with advanced dementia. Alzheimer Dis Assoc Disord. 2006 Oct-Dec;20(4):283-90. doi: 10.1097/01.wad.0000213854.04861.cc. PMID 17132974
- [Background] Boerlage AA, van Dijk M, Stronks DL, de Wit R, van der Rijt CC. Pain prevalence and characteristics in three Dutch residential homes. Eur J Pain. 2008 Oct;12(7):910-6. doi: 10.1016/j.ejpain.2007.12.014. Epub 2008 Feb 11. PMID 18267371
- [Background] Cook AJ. Cognitive-behavioral pain management for elderly nursing home residents. J Gerontol B Psychol Sci Soc Sci. 1998 Jan;53(1):P51-9. doi: 10.1093/geronb/53b.1.p51. PMID 9469172
- [Background] D'Astolfo CJ, Humphreys BK. A record review of reported musculoskeletal pain in an Ontario long term care facility. BMC Geriatr. 2006 Mar 23;6:5. doi: 10.1186/1471-2318-6-5. PMID 16556306
- [Background] Damian J, Valderrama-Gama E, Rodriguez-Artalejo F, Martin-Moreno JM. [Health and functional status among elderly individuals living in nursing homes in Madrid]. Gac Sanit. 2004 Jul-Aug;18(4):268-74. doi: 10.1016/s0213-9111(04)72013-0. Spanish. PMID 15324637
- [Background] Decker SA, Culp KR, Cacchione PZ. Evaluation of musculoskeletal pain management practices in rural nursing homes compared with evidence-based criteria. Pain Manag Nurs. 2009 Jun;10(2):58-64. doi: 10.1016/j.pmn.2008.02.008. Epub 2008 Nov 7. PMID 19481044
- [Background] Ferrell BA, Ferrell BR, Osterweil D. Pain in the nursing home. J Am Geriatr Soc. 1990 Apr;38(4):409-14. doi: 10.1111/j.1532-5415.1990.tb03538.x. PMID 2109765
- [Background] U.H. Finne-Soveri, G. Ljunggren, M. Schroll, P.V. Jonsson, I. Hjaltadottir, K. El Kholy, R.S. Tilvis, Pain and its association with disability in institutional long-term care in four Nordic countries, Canadian Journal on Aging 19(SUPPL. 2) (2000) 38-49.
- [Background] Fisher SE, Burgio LD, Thorn BE, Allen-Burge R, Gerstle J, Roth DL, Allen SJ. Pain assessment and management in cognitively impaired nursing home residents: association of certified nursing assistant pain report, Minimum Data Set pain report, and analgesic medication use. J Am Geriatr Soc. 2002 Jan;50(1):152-6. doi: 10.1046/j.1532-5415.2002.50021.x. PMID 12028260
- [Background] Gill TK, Caughey GE, Wesselingh S, Inacio MC. Impact of musculoskeletal conditions among those in residential aged care in Australia. Australas J Ageing. 2022 Mar;41(1):e41-e49. doi: 10.1111/ajag.13001. Epub 2021 Oct 5. PMID 34611957
- [Background] Gerber AM, Botes R, Mostert A, Vorster A, Buskens E. A cohort study of elderly people in Bloemfontein, South Africa, to determine health-related quality of life and functional abilities. S Afr Med J. 2016 Feb 4;106(3):298-301. doi: 10.7196/SAMJ.2016.v106i3.10171. PMID 26915946
- [Background] Grimby C, Fastbom J, Forsell Y, Thorslund M, Claesson CB, Winblad B. Musculoskeletal pain and analgesic therapy in a very old population. Arch Gerontol Geriatr. 1999 Jul-Aug;29(1):29-43. doi: 10.1016/s0167-4943(99)00021-7. PMID 15374075
- [Background] Guccione AA, Meenan RF, Anderson JJ. Arthritis in nursing home residents. A validation of its prevalence and examination of its impact on institutionalization and functional status. Arthritis Rheum. 1989 Dec;32(12):1546-53. doi: 10.1002/anr.1780321208. PMID 2597209
- [Background] Hillen JB, Vitry A, Caughey GE. Disease burden, comorbidity and geriatric syndromes in the Australian aged care population. Australas J Ageing. 2017 Jun;36(2):E14-E19. doi: 10.1111/ajag.12411. Epub 2017 Apr 11. PMID 28401631
- [Background] Hsieh SW, Huang LC, Hsieh TJ, Lin CF, Hsu CC, Yang YH. Behavioral and psychological symptoms in institutional residents with dementia in Taiwan. Geriatr Gerontol Int. 2021 Aug;21(8):718-724. doi: 10.1111/ggi.14220. Epub 2021 Jun 28. PMID 34184383
- [Background] Jerez-Roig J, Souza DL, Andrade FL, Lima BF Filho, Medeiros RJ, Oliveira NP, Cabral SM Neto, Lima KC. Self-perceived health in institutionalized elderly. Cien Saude Colet. 2016 Nov;21(11):3367-3375. doi: 10.1590/1413-812320152111.15562015. English, Portuguese. PMID 27828570
- [Background] Kalideen L, Van Wyk JM, Govender P. Demographic and clinical profiles of residents in long-term care facilities in South Africa: A cross-sectional survey. Afr J Prim Health Care Fam Med. 2022 Mar 18;14(1):e1-e9. doi: 10.4102/phcfm.v14i1.3131. PMID 35384684
- [Background] R. Karmel, D. Gibson, P. Anderson, Y. Wells, S. Duckett, Care trajectories through community and residential aged care services: disease effects, Ageing & Society 32 (2012) 1428-1445.
- [Background] Lapane KL, Quilliam BJ, Chow W, Kim M. The association between pain and measures of well-being among nursing home residents. J Am Med Dir Assoc. 2012 May;13(4):344-9. doi: 10.1016/j.jamda.2011.01.007. Epub 2011 Mar 23. PMID 21450246
- [Background] Lind KE, Raban MZ, Brett L, Jorgensen ML, Georgiou A, Westbrook JI. Measuring the prevalence of 60 health conditions in older Australians in residential aged care with electronic health records: a retrospective dynamic cohort study. Popul Health Metr. 2020 Oct 8;18(1):25. doi: 10.1186/s12963-020-00234-z. PMID 33032628
- [Background] Luque Ramos A, Albrecht K, Zink A, Hoffmann F. Rheumatologic care of nursing home residents with rheumatoid arthritis: a comparison of the year before and after nursing home admission. Rheumatol Int. 2017 Dec;37(12):2059-2064. doi: 10.1007/s00296-017-3791-5. Epub 2017 Aug 18. PMID 28821941
- [Background] A. Marques, V. Rocha, M. Pinto, L. Sousa, D. Figueiredo, Comorbidities and medication intake among people with dementia living in long-term care facilities, Revista Portuguesa de Saude Publica 33(1) (2015) 42-48.
- [Background] Martinez-Gallardo Prieto L, Hermida Galindo LF, D'hyver de Las Deses C. [Prevalence of foot conditions in a geriatric population and their impact on mobility, gait and tendency to falls]. Rev Esp Geriatr Gerontol. 2012 Jan-Feb;47(1):19-22. doi: 10.1016/j.regg.2011.05.004. Epub 2011 Oct 14. Spanish. PMID 22000071
- [Background] Monroe T, Carter M, Parish A. A case study using the beers list criteria to compare prescribing by family practitioners and geriatric specialists in a rural nursing home. Geriatr Nurs. 2011 Sep-Oct;32(5):350-6. doi: 10.1016/j.gerinurse.2011.07.003. PMID 21962885
- [Background] Moore KL, Boscardin WJ, Steinman MA, Schwartz JB. Age and sex variation in prevalence of chronic medical conditions in older residents of U.S. nursing homes. J Am Geriatr Soc. 2012 Apr;60(4):756-64. doi: 10.1111/j.1532-5415.2012.03909.x. Epub 2012 Mar 29. PMID 22463062
- [Background] Ng R, Lane N, Tanuseputro P, Mojaverian N, Talarico R, Wodchis WP, Bronskill SE, Hsu AT. Increasing Complexity of New Nursing Home Residents in Ontario, Canada: A Serial Cross-Sectional Study. J Am Geriatr Soc. 2020 Jun;68(6):1293-1300. doi: 10.1111/jgs.16394. Epub 2020 Mar 2. PMID 32119121
- [Background] Nguyen AD, Lind KE, Day RO, Georgiou A, Westbrook JI. A profile of health status and demographics of aged care facility residents with gout. Australas J Ageing. 2020 Mar;39(1):e153-e161. doi: 10.1111/ajag.12716. Epub 2019 Aug 21. PMID 31433129
- [Background] Peng LN, Lin MH, Lai HY, Hwang SJ, Chen LK, Lan CF. Pain and health-care utilization among older men in a veterans care home. Arch Gerontol Geriatr. 2009 Dec;49 Suppl 2:S13-6. doi: 10.1016/S0167-4943(09)70006-8. PMID 20005419
- [Background] Proctor WR, Hirdes JP. Pain and cognitive status among nursing home residents in Canada. Pain Res Manag. 2001 Fall;6(3):119-25. doi: 10.1155/2001/978130. PMID 11854774
- [Background] Van Rensbergen G, Nawrot T. Medical conditions of nursing home admissions. BMC Geriatr. 2010 Jul 14;10:46. doi: 10.1186/1471-2318-10-46. PMID 20630079
- [Background] Sawyer P, Lillis JP, Bodner EV, Allman RM. Substantial daily pain among nursing home residents. J Am Med Dir Assoc. 2007 Mar;8(3):158-65. doi: 10.1016/j.jamda.2006.12.030. PMID 17349944
- [Background] A.K. Sigurdardottir, K. Olafsson, R.H. Arnardottir, I. Hjaltadottir, Health status and functional profile at admission to nursing homes a population based study over the years 2003-2014: Comparison between people with and without diabetes, Journal of Gerontology and Geriatrics 66(3) (2018) 134-141.
- [Background] Takai Y, Yamamoto-Mitani N, Fukahori H, Kobayashi S, Chiba Y. Nursing ward managers' perceptions of pain prevalence at the aged-care facilities in Japan: a nationwide survey. Pain Manag Nurs. 2013 Sep;14(3):e59-66. doi: 10.1016/j.pmn.2011.04.004. Epub 2011 Jun 17. PMID 23972872
- [Background] Tansug M, Kahraman T, Genc A. Differences in Pain Characteristics and Functional Associations between Nursing Home Residents and Community-Dwelling Older Adults: A Cross-Sectional Study. Ann Geriatr Med Res. 2021 Sep;25(3):187-196. doi: 10.4235/agmr.21.0066. Epub 2021 Aug 26. PMID 34433255
- [Background] Torvik K, Kaasa S, Kirkevold O, Rustoen T. Pain and quality of life among residents of Norwegian nursing homes. Pain Manag Nurs. 2010 Mar;11(1):35-44. doi: 10.1016/j.pmn.2009.01.001. Epub 2009 Dec 30. PMID 20207326
- [Background] Tsai YF, Tsai HH, Lai YH, Chu TL. Pain prevalence, experiences and management strategies among the elderly in taiwanese nursing homes. J Pain Symptom Manage. 2004 Dec;28(6):579-84. doi: 10.1016/j.jpainsymman.2004.03.007. PMID 15589082
- [Background] Tse MM, Pun SP, Benzie IF. Pain relief strategies used by older people with chronic pain: an exploratory survey for planning patient-centred intervention. J Clin Nurs. 2005 Mar;14(3):315-20. doi: 10.1111/j.1365-2702.2004.00976.x. PMID 15707441
- [Background] Veal F, Williams M, Bereznicki L, Cummings E, Winzenberg T. A retrospective review of pain management in Tasmanian residential aged care facilities. BJGP Open. 2019 Mar 6;3(1):bjgpopen18X101629. doi: 10.3399/bjgpopen18X101629. eCollection 2019 Apr. PMID 31049410
- [Background] Zanocchi M, Maero B, Nicola E, Martinelli E, Luppino A, Gonella M, Gariglio F, Fissore L, Bardelli B, Obialero R, Molaschi M. Chronic pain in a sample of nursing home residents: prevalence, characteristics, influence on quality of life (QoL). Arch Gerontol Geriatr. 2008 Jul-Aug;47(1):121-8. doi: 10.1016/j.archger.2007.07.003. Epub 2007 Nov 19. PMID 18006088
- [Background] Zarowitz BJ, O'Shea TE. Demographic and clinical profile of nursing facility residents with gout. Consult Pharm. 2013 Jun;28(6):370-82. doi: 10.4140/TCP.n.2013.370. PMID 23748125